CLINICAL TRIAL: NCT02882880
Title: The Treatment of Sleep Bruxism With the Luco Hybrid OSA Appliance
Brief Title: Treatment Sleep Bruxism With the Luco Hybrid OSA Appliance
Acronym: LucoHybrid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luco Hybrid OSA Appliance Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Ken Luco, Principal Investigator, Luco Hybrid OSA Appliance Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Lucohybridosa
Record Dates: First submitted 2016-08-21; First posted 2016-08-30 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Sleep Bruxism; Tension Headache; Migraine Headache
MeSH Terms: conditions — Sleep Bruxism; Tension-Type Headache; Migraine Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Started (Other): Intervention: Treatment with the Luco Hybrid OSA Appliance (LHOA) Group 1, fitted with LHOA Group 2: LHOA removed for 48 hours
  Interventions: Device: The Luco Hybrid OSA Appliance
- Completed (Active Comparator): Intervention: The LUco Hybrid OSA APpliance The subjects that actually completed the study in both groups. Group 1 n = 32, in Group 2 n=19
  Interventions: Device: The Luco Hybrid OSA Appliance

INTERVENTIONS:
Device: The Luco Hybrid OSA Appliance — Group 1, initial treatment with the device, reassessed at 14 and 60 days, Group 2, removal of the treatment for 48 hours, to determine if relapse occurs, retested at 60 days with the device (recovery from intervention).
  Other Names: Mandibular advancement appliance

SUMMARY:
To determine the effectiveness of the Luco Hybrid OSA Appliance in the treatment of sleep bruxism and to aid in the treatment of associated tension/migraine type headaches in adults.

DETAILED DESCRIPTION:
51 subjects were selected and separated into two groups: those new to the treatment (Group 1)and those who had been in treatment for more than 1 year (Group 2). There were 32 participants in group 1 and 19 in group 2. mean age for Group 1 was 41.7 and Group 2 was 50.5. The age range for Group 1 was 21 to 66 and in Group 2 34 to 73.

Group 1 subjects were fitted with a Luco hybrid OSA appliance (LHOA). They were followed over a 14 day period with adjustments made to the device as required. The second study [milestone] was completed at that time.

Group 2 subjects, who had previously been in treatment with the device for and mean of 4.1 years, had an initial study with the device and a second study following 48 hours without the device.

Both groups were studied again at 60 days and results compared.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age (adult)
* capable of giving informed consent
* met the AASM criteria for sleep bruxism
* had sound dentition
* did not have active obstructive sleep apnea(OSA)/upper airway resistance syndrome (UARS)

Exclusion Criteria:

* younger than 18
* incapable of informed consent
* did not meet the AASM criteria for sleep bruxism
* discovered OSA or UARS in the initial study
* did not have sound dentition (active caries, periodontal disease, inadequate number of teeth
* had obstructive sleep apnea/UARS
* did not complete the study
* completed the study but did not complete all aspects of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-07; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Response to treatment with the Luco Hybrid OSA Appliance | 60 days
  Clinical examination, sleep study and visual analog scale. Clinical examination of the subject's musculature, temporomandibular joints (TMJ), and measurement of the range of mandibular movements. The home sleep study (HSS) measured the number and duration of sleep bruxism events as well as the heart rate associated with these events. The visual analog scale (VAS) recorded the patient's response regarding TMJ pain on waking and later in the day, jaw muscle pain on waking and later in the day, tooth sensitivity to temperature extremes, tension/migraine type headaches on waking and later in the day and neck/shoulder pain on waking and later in the day.
  HSS scoring according to the American Academy of Sleep Medicine's "Manual for the Scoring of Sleep and Associated Events" for sleep bruxism.

CONTACTS AND LOCATIONS:
Overall Officials: Ken J Luco, DDS, BSc, Principal Investigator — Luco Hybrid OSA Appliance Inc.
Locations (1):
- Dr. K. Luco Dentistry Professional Corporation, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klasser GD, Greene CS, Lavigne GJ. Oral appliances and the management of sleep bruxism in adults: a century of clinical applications and search for mechanisms. Int J Prosthodont. 2010 Sep-Oct;23(5):453-62. PMID 20859563
- [Background] Raphael KG, Santiago V, Lobbezoo F. Is bruxism a disorder or a behaviour? Rethinking the international consensus on defining and grading of bruxism. J Oral Rehabil. 2016 Oct;43(10):791-8. doi: 10.1111/joor.12413. Epub 2016 Jun 10. PMID 27283599
- [Background] Tavares LM, da Silva Parente Macedo LC, Duarte CM, de Goffredo Filho GS, de Souza Tesch R. Cross-sectional study of anxiety symptoms and self-report of awake and sleep bruxism in female TMD patients. Cranio. 2016 Nov;34(6):378-381. doi: 10.1080/08869634.2016.1163806. Epub 2016 Apr 20. PMID 27097685
- [Background] Gomes CAFP, El-Hage Y, Amaral AP, Herpich CM, Politti F, Kalil-Bussadori S, Gonzalez TO, Biasotto-Gonzalez DA. Effects of Massage Therapy and Occlusal Splint Usage on Quality of Life and Pain in Individuals with Sleep Bruxism: A Randomized Controlled Trial. J Jpn Phys Ther Assoc. 2015;18(1):1-6. doi: 10.1298/jjpta.Vol18_001. PMID 26733760
- [Background] Dharmadhikari S, Romito LM, Dzemidzic M, Dydak U, Xu J, Bodkin CL, Manchanda S, Byrd KE. GABA and glutamate levels in occlusal splint-wearing males with possible bruxism. Arch Oral Biol. 2015 Jul;60(7):1021-9. doi: 10.1016/j.archoralbio.2015.03.006. Epub 2015 Mar 28. PMID 25889171
- [Background] Hesselbacher S, Subramanian S, Rao S, Casturi L, Surani S. Self-reported sleep bruxism and nocturnal gastroesophageal reflux disease in patients with obstructive sleep apnea: relationship to gender and ethnicity. Open Respir Med J. 2014 Oct 22;8:34-40. doi: 10.2174/1874306401408010034. eCollection 2014. PMID 25352924
- [Result] Carra MC, Huynh N, Fleury B, Lavigne G. Overview on Sleep Bruxism for Sleep Medicine Clinicians. Sleep Med Clin. 2015 Sep;10(3):375-84, xvi. doi: 10.1016/j.jsmc.2015.05.005. Epub 2015 Jul 8. PMID 26329448
- [Result] Mayer P, Heinzer R, Lavigne G. Sleep Bruxism in Respiratory Medicine Practice. Chest. 2016 Jan;149(1):262-71. doi: 10.1378/chest.15-0822. Epub 2016 Jan 6. PMID 26225899
- [Result] Klasser GD, Rei N, Lavigne GJ. Sleep bruxism etiology: the evolution of a changing paradigm. J Can Dent Assoc. 2015;81:f2. PMID 25633110
- [Result] Saito M, Yamaguchi T, Mikami S, Watanabe K, Gotouda A, Okada K, Hishikawa R, Shibuya E, Lavigne G. Temporal association between sleep apnea-hypopnea and sleep bruxism events. J Sleep Res. 2013 Nov 4. doi: 10.1111/jsr.12099. Online ahead of print. PMID 24635459
- [Result] Hasegawa Y, Lavigne G, Rompre P, Kato T, Urade M, Huynh N. Is there a first night effect on sleep bruxism? A sleep laboratory study. J Clin Sleep Med. 2013 Nov 15;9(11):1139-45. doi: 10.5664/jcsm.3152. PMID 24235894
- [Result] Abe S, Gagnon JF, Montplaisir JY, Postuma RB, Rompre PH, Huynh NT, Kato T, Kawano F, Lavigne GJ. Sleep bruxism and oromandibular myoclonus in rapid eye movement sleep behavior disorder: a preliminary report. Sleep Med. 2013 Oct;14(10):1024-30. doi: 10.1016/j.sleep.2013.04.021. Epub 2013 Aug 15. PMID 23953215
- [Result] Raphael KG, Sirois DA, Janal MN, Wigren PE, Dubrovsky B, Nemelivsky LV, Klausner JJ, Krieger AC, Lavigne GJ. Sleep bruxism and myofascial temporomandibular disorders: a laboratory-based polysomnographic investigation. J Am Dent Assoc. 2012 Nov;143(11):1223-31. doi: 10.14219/jada.archive.2012.0068. PMID 23115152
- [Result] Carra MC, Huynh N, Lavigne G. Sleep bruxism: a comprehensive overview for the dental clinician interested in sleep medicine. Dent Clin North Am. 2012 Apr;56(2):387-413. doi: 10.1016/j.cden.2012.01.003. PMID 22480810
- [Result] Nashed A, Lanfranchi P, Rompre P, Carra MC, Mayer P, Colombo R, Huynh N, Lavigne G. Sleep bruxism is associated with a rise in arterial blood pressure. Sleep. 2012 Apr 1;35(4):529-36. doi: 10.5665/sleep.1740. PMID 22467991
- [Result] Franco L, Rompre PH, de Grandmont P, Abe S, Lavigne GJ. A mandibular advancement appliance reduces pain and rhythmic masticatory muscle activity in patients with morning headache. J Orofac Pain. 2011 Summer;25(3):240-9. PMID 21837291
- [Result] Lavigne G, Palla S. Transient morning headache: recognizing the role of sleep bruxism and sleep-disordered breathing. J Am Dent Assoc. 2010 Mar;141(3):297-9. doi: 10.14219/jada.archive.2010.0163. No abstract available. PMID 20194385
- [Result] Landry-Schonbeck A, de Grandmont P, Rompre PH, Lavigne GJ. Effect of an adjustable mandibular advancement appliance on sleep bruxism: a crossover sleep laboratory study. Int J Prosthodont. 2009 May-Jun;22(3):251-9. PMID 19548407
- [Result] Huynh NT, Rompre PH, Montplaisir JY, Manzini C, Okura K, Lavigne GJ. Comparison of various treatments for sleep bruxism using determinants of number needed to treat and effect size. Int J Prosthodont. 2006 Sep-Oct;19(5):435-41. PMID 17323720
- [Result] Landry ML, Rompre PH, Manzini C, Guitard F, de Grandmont P, Lavigne GJ. Reduction of sleep bruxism using a mandibular advancement device: an experimental controlled study. Int J Prosthodont. 2006 Nov-Dec;19(6):549-56. PMID 17165292
- [Result] Huynh N, Lavigne GJ, Lanfranchi PA, Montplaisir JY, de Champlain J. The effect of 2 sympatholytic medications--propranolol and clonidine--on sleep bruxism: experimental randomized controlled studies. Sleep. 2006 Mar;29(3):307-16. doi: 10.1093/sleep/29.3.307. PMID 16553016
- [Result] Lavigne G, Kato T. Usual and unusual orofacial motor activities associated with tooth wear. Int J Prosthodont. 2005 Jul-Aug;18(4):291-2. No abstract available. PMID 16052775
- [Result] Miyawaki S, Lavigne GJ, Pierre M, Guitard F, Montplaisir JY, Kato T. Association between sleep bruxism, swallowing-related laryngeal movement, and sleep positions. Sleep. 2003 Jun 15;26(4):461-5. PMID 12841373
- [Result] Ohmure H, Kanematsu-Hashimoto K, Nagayama K, Taguchi H, Ido A, Tominaga K, Arakawa T, Miyawaki S. Evaluation of a Proton Pump Inhibitor for Sleep Bruxism: A Randomized Clinical Trial. J Dent Res. 2016 Dec;95(13):1479-1486. doi: 10.1177/0022034516662245. Epub 2016 Jul 29. PMID 27474257
- [Result] Cahlin BJ, Hedner J, Dahlstrom L. A randomised, open-label, crossover study of the dopamine agonist, pramipexole, in patients with sleep bruxism. J Sleep Res. 2017 Feb;26(1):64-72. doi: 10.1111/jsr.12440. Epub 2016 Jul 17. PMID 27426276
- [Result] Solanki N, Singh BP, Chand P, Siddharth R, Arya D, Kumar L, Tripathi S, Jivanani H, Dubey A. Effect of mandibular advancement device on sleep bruxism score and sleep quality. J Prosthet Dent. 2017 Jan;117(1):67-72. doi: 10.1016/j.prosdent.2016.04.009. Epub 2016 Jul 14. PMID 27422230
- [Result] Okura K, Shigemoto S, Suzuki Y, Noguchi N, Omoto K, Abe S, Matsuka Y. Mandibular movement during sleep bruxism associated with current tooth attrition. J Prosthodont Res. 2017 Jan;61(1):87-95. doi: 10.1016/j.jpor.2016.06.003. Epub 2016 Jun 25. PMID 27354030
- [Result] Zhou WN, Fu HY, Du YF, Sun JH, Zhang JL, Wang C, Svensson P, Wang KL. Short-term effects of repetitive transcranial magnetic stimulation on sleep bruxism - a pilot study. Int J Oral Sci. 2016 Mar 30;8(1):61-5. doi: 10.1038/ijos.2015.35. PMID 27025267
- [Result] Guaita M, Hogl B. Current Treatments of Bruxism. Curr Treat Options Neurol. 2016 Feb;18(2):10. doi: 10.1007/s11940-016-0396-3. PMID 26897026
- [Result] Castrillon EE, Ou KL, Wang K, Zhang J, Zhou X, Svensson P. Sleep bruxism: an updated review of an old problem. Acta Odontol Scand. 2016 Jul;74(5):328-34. doi: 10.3109/00016357.2015.1125943. Epub 2016 Jan 12. PMID 26758348
- [Result] Minakuchi H, Sogawa C, Miki H, Hara ES, Maekawa K, Sogawa N, Kitayama S, Matsuka Y, Clark GT, Kuboki T. Sleep bruxism frequency and platelet serotonin transporter activities in young adult subjects. Sleep Breath. 2016 Mar;20(1):271-6. doi: 10.1007/s11325-015-1281-0. Epub 2015 Nov 2. PMID 26527205
- [Result] Malcmacher L. Ensuring Restorative Success With Bruxism Testing. Dent Today. 2015 Jul;34(7):131-3. No abstract available. PMID 26285347
- [Result] Malcmacher L. Bruxism--Are You Helping or Hurting Your Patients? J N J Dent Assoc. 2015 Winter;86(1):14-6. No abstract available. PMID 26215023
- [Result] Kostrzewa-Janicka J, Jurkowski P, Zycinska K, Przybylowska D, Mierzwinska-Nastalska E. Sleep-Related Breathing Disorders and Bruxism. Adv Exp Med Biol. 2015;873:9-14. doi: 10.1007/5584_2015_151. PMID 26022906
- [Result] Gu W, Yang J, Zhang F, Yin X, Wei X, Wang C. Efficacy of biofeedback therapy via a mini wireless device on sleep bruxism contrasted with occlusal splint: a pilot study. J Biomed Res. 2015 Apr;29(2):160-8. doi: 10.7555/JBR.28.20130145. Epub 2014 Nov 18. PMID 25859272
- [Result] Gomes CA, El Hage Y, Amaral AP, Politti F, Biasotto-Gonzalez DA. Effects of massage therapy and occlusal splint therapy on electromyographic activity and the intensity of signs and symptoms in individuals with temporomandibular disorder and sleep bruxism: a randomized clinical trial. Chiropr Man Therap. 2014 Dec 15;22(1):43. doi: 10.1186/s12998-014-0043-6. eCollection 2014. PMID 25512839
- [Result] Stark CD, Stark RJ. Sleep and chronic daily headache. Curr Pain Headache Rep. 2015 Jan;19(1):468. doi: 10.1007/s11916-014-0468-6. PMID 25416461
- [Result] Matsumoto H, Tsukiyama Y, Kuwatsuru R, Koyano K. The effect of intermittent use of occlusal splint devices on sleep bruxism: a 4-week observation with a portable electromyographic recording device. J Oral Rehabil. 2015 Apr;42(4):251-8. doi: 10.1111/joor.12251. Epub 2014 Nov 1. PMID 25363423
- [Result] Malcmacher L. Are you prescribing bruxism appliances? Dent Today. 2014 Sep;33(9):126-9. No abstract available. PMID 25283030
- [Result] Yamaguchi K, Ishiura Y, Tanaka S, Baba K. Influence of the rigidity of a provisional restoration supported on four immediately loaded implants in the edentulous maxilla on biomechanical bone-implant interactions under simulated bruxism conditions: a three-dimensional finite element analysis. Int J Prosthodont. 2014 Sep-Oct;27(5):442-50. doi: 10.11607/ijp.3857. PMID 25191887
- [Result] Porporatti AL, Costa YM, Conti PC, Bonjardim LR, Calderon Pdos S. Primary headaches interfere with the efficacy of temporomandibular disorders management. J Appl Oral Sci. 2015 Mar-Apr;23(2):129-34. doi: 10.1590/1678-775720130557. Epub 2014 Jul 4. PMID 25004051
- [Result] Sjoholm T, Kauko T, Kemppainen P, Rauhala E. Long-term use of occlusal appliance has impact on sleep structure. J Oral Rehabil. 2014 Nov;41(11):795-800. doi: 10.1111/joor.12201. Epub 2014 Jun 18. PMID 24942041
- [Result] Chate R. Summary of: Over-the-counter (OTC) bruxism splints available on the Internet. Br Dent J. 2014 Jun 13;216(11):642-3. doi: 10.1038/sj.bdj.2014.480. No abstract available. PMID 24923944
- [Result] de-la-Hoz JL. Sleep bruxism: review and update for the restorative dentist. Alpha Omegan. 2013 Spring-Summer;106(1-2):23-8. PMID 24864394
- [Result] Karakis D, Dogan A, Bek B. Evaluation of the effect of two different occlusal splints on maximum occlusal force in patients with sleep bruxism: a pilot study. J Adv Prosthodont. 2014 Apr;6(2):103-8. doi: 10.4047/jap.2014.6.2.103. Epub 2014 Apr 22. PMID 24843394
- [Result] Mainieri VC, Saueressig AC, Fagondes SC, Teixeira ER, Rehm DD, Grossi ML. Analysis of the effects of a mandibular advancement device on sleep bruxism using polysomnography, the BiteStrip, the sleep assessment questionnaire, and occlusal force. Int J Prosthodont. 2014 Mar-Apr;27(2):119-26. doi: 10.11607/ijp.3675. PMID 24596907
- [Result] Sumiya M, Mizumori T, Kobayashi Y, Inano S, Yatani H. Suppression of sleep bruxism: effect of electrical stimulation of the masseter muscle triggered by heart rate elevation. Int J Prosthodont. 2014 Jan-Feb;27(1):80-6. doi: 10.11607/ijp.3330. PMID 24392483
- [Result] Huang H, Song YH, Wang JJ, Guo Q, Liu WC. Excitability of the central masticatory pathways in patients with sleep bruxism. Neurosci Lett. 2014 Jan 13;558:82-6. doi: 10.1016/j.neulet.2013.11.014. Epub 2013 Nov 20. PMID 24269982
- [Result] Saletu B, Anderer P, Saletu-Zyhlarz GM. Recent advances in sleep research. Psychiatr Danub. 2013 Dec;25(4):426-34. PMID 24247058
- [Result] Lin XL, Tang SY. Sodium valproate may be a treatment for sleep bruxism. J Child Adolesc Psychopharmacol. 2013 Nov;23(9):636-7. doi: 10.1089/cap.2013.0015. Epub 2013 Oct 29. No abstract available. PMID 24168714
- [Result] Aqueveque P, Pino E, Lopez R. Electrical stimulation device as possible treatment for nocturnal bruxism: preliminary results. Annu Int Conf IEEE Eng Med Biol Soc. 2013;2013:3571-3. doi: 10.1109/EMBC.2013.6610314. PMID 24110501
- [Result] Wang LF, Long H, Deng M, Xu H, Fang J, Fan Y, Bai D, Han XL. Biofeedback treatment for sleep bruxism: a systematic review. Sleep Breath. 2014 May;18(2):235-42. doi: 10.1007/s11325-013-0871-y. Epub 2013 Jun 12. PMID 23756884
- [Result] Carra MC, Huynh NT, El-Khatib H, Remise C, Lavigne GJ. Sleep bruxism, snoring, and headaches in adolescents: short-term effects of a mandibular advancement appliance. Sleep Med. 2013 Jul;14(7):656-61. doi: 10.1016/j.sleep.2013.03.009. Epub 2013 May 2. PMID 23643652
- [Result] Dowd ET. Nocturnal bruxism and hypnotherapy: a case study. Int J Clin Exp Hypn. 2013;61(2):205-18. doi: 10.1080/00207144.2013.753832. PMID 23427844
- [Result] Silber MH. Sleep-related movement disorders. Continuum (Minneap Minn). 2013 Feb;19(1 Sleep Disorders):170-84. doi: 10.1212/01.CON.0000427207.13553.68. PMID 23385700